CLINICAL TRIAL: NCT01111344
Title: Efficacy of Glizigen-Viudid in the Treatment of External Anogenital Warts in Children and Adolescents.
Brief Title: Glizigen-Viudid-External Anogenital Warts in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-1002-CU
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: External Anogenital Warts
Keywords: Dietary supplement; Anogenital warts; Viusid; Glizigen
MeSH Terms: conditions — Condylomata Acuminata | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glizigen + Viusid (Experimental)
  Interventions: Dietary Supplement: Glizigen + Viusid
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glizigen + Viusid — Glizigen (spray, 60 mL bottle with applicator): Dosage commensurate with surface (up to a maximum of 10 cm2) to be treated. From 3 to 5 ambulatory applications (One nebulization corresponds to 2 short pulses).
  * 1 to 3.9 cm2 ______________3 daily applications
  * 4 to 6.9 cm2 ______________4 daily applications
  * 7 to 10 cm2 ______________5 daily applications Treatment will last from 5 days to 8 weeks according to clinical improvement.
  Viusid (Syrop, 500 mL flask): 12.5 ml every 8 hours for 12 weeks. Viusid syrop should be dissolved in water, fruit juice or milk before ingestion.
  Arms: Glizigen + Viusid
Dietary Supplement: Placebo — Placebo Glizipen (spray, 60 mL bottle with applicator): Dosage commensurate with surface (up to a maximum of 10 cm2) to be treated. From 3 to 5 ambulatory applications (One nebulization corresponds to 2 short pulses).
  * 1 to 3.9 cm2 ______________3 daily applications
  * 4 to 6.9 cm2 ______________4 daily applications
  * 7 to 10 cm2 ______________5 daily applications Treatment will last from 5 days to 8 weeks according to clinical improvement.
  Placebo Viusid (Syrop, 500 mL flask): 12.5 ml every 8 hours for 12 weeks. Viusid syrop should be dissolved in water, fruit juice or milk before ingestion.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy of Glizigen and Viusid administration in the treatment of external anogenital warts in children and adolescents. The duration of this double-blind placebo controlled phase 3 clinical trial will be 12 weeks. The estimated number of persons to be recruited and randomized for the study is 76. Variables to be assessed will be: time to disappearance of lesions, reduction of the number of lesions and change in the aspect of lesions.

ELIGIBILITY:
Inclusion Criteria:

* No previous treatment for anogenital warts
* Negative serology for HB and HIV.
* Signed informed consent.

Exclusion Criteria:

* Pregnancy
* Treatment with steroids, immune-suppressors, immune-modulators or local or systemic antiviral drugs.
* Hypersensitivity to Glizigen or Viusid:

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Time to lesion regression | 12 weeks
  Excellent: Lesion regression before 2 weeks of treatment Good: Lesion regression between 2-5 weeks of treatment Poor: Lesion regression between 5-8 weeks of treatment Bad: No lesion regression after 8 weeks of treatment.

SECONDARY OUTCOMES:
Occurrence of adverse effects within the 12 week treatment period | 12 weeks
Reduction in the number of lesions | 12 weeks
  Excellent: Regression in more than 75% of lesions Good: Regression in 50-75% of lesions Poor: Regression in 25-50% of lesions Bad: Regression in less than 25% of lesions.
Lesion aspect | 12 weeks
  Excellent: Lesion regression Poor: Aspect changes from papilloma shaped to flat shaped lesion. Bad: No change in aspect or change from flat shaped to papilloma shaped lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Edelisa Moredo Romo, MD, Principal Investigator — Pediatric Hospital "Dr. Juan Manuel Márquez.
Locations (1):
- Pediatric Hospital "Dr. Juan Manuel Márquez"., Havana, La Habana, Cuba